CLINICAL TRIAL: NCT01474577
Title: Prognostic Value of Rb-82 PET Myocardial Perfusion Imaging
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-150
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2016-11

CONDITIONS: Cardiac Health
Keywords: stress test; cardiac issues; Rb-82 PET Myocardial Perfusion Imaging; 11-150; one or more 82Rb myocardial perfusion stress tests
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- pts who have had Rb-82 PET myocardial perfusion imaging: Eligible patients will have had Rb-82 PET myocardial perfusion imaging at MSKCC, 2008 - 2011. Patients will complete one questionnaire over the phone.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Patients will complete one questionnaire over the phone. We will ask patients to describe their cardiac history since Rb-82 PET (chest pain, shortness of breath, cardiac catheterization, and heart attack). This information will be correlated to the scan results and other relevant information in the patient's medical record.

SUMMARY:
The physician would like to see if nuclear cardiac stress tests can predict cardiac health. For example, if a patient has an abnormal stress test, is he or she more likely to have cardiac problems in the future?

ELIGIBILITY:
Inclusion Criteria:

* Patient > or = to 18 years of age
* Registered patient at MSKCC
* Patient with one or more 82Rb myocardial perfusion stress tests performed at MSKCC, 2008-2011

Exclusion Criteria:

* Patient is unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with one or more 82Rb myocardial perfusion stress tests performed at MSKCC, 2008-2011.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2011-11-08 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
correlate scan findings with clinical outcomes | 1 year
  Patients will complete one questionnaire over the phone.

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schöder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/